CLINICAL TRIAL: NCT00476177
Title: Infusion of Donor Dendritic Cells and Donor Lymphocytes in Patients With Relapsed Hematologic Malignancies After Allogenic Transplant
Brief Title: Donor Dendritic Cells And Donor Lymphocytes in Patients With Relapsed Hematologic Malignancies After Allogeneic Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edwin P. Alyea, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-003
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Hematologic Malignancy
Keywords: DC; DLI; graft vs. host disease; GVHD
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Infusion of donor dendritic cells — Given in the outpatient setting
Biological: Infusion of donor lymphocytes — Given in outpatient setting

SUMMARY:
The purpose of this study is to test the safety of adding donor dendritic cells to donor lymphocyte infusions, and to determine the type and severity of any side effects associated with this addition. Previously patients with hematologic malignancies who relapsed after transplant have been given infusions of donor white blood cells (donor lymphocyte infusion, DLI) as a way to boost their immune function and fight disease. Although DLI has led to cancer regression in some patients, the overall response rate using DLI alone is low, and unfortunately, rarely lasting. Researchers have discovered a new subset of blood cells, called dendritic cells (DC), which are crucial partners to lymphocytes in generating an immune response. We believe that the infusion of DC together with DLI may improve the ability of the donor lymphocytes to recognize and kill cancer cells.

DETAILED DESCRIPTION:
* Since we are looking for the highest dose of donor dendritic cells that can be administered safely with DLI patients after allogeneic stem cell transplant, not everyone who participates in this study will be receiving the same number of dendritic cells.
* The study procedure can be divided into 3 phases: 1) Pre-infusion evaluation, 2) Cell collections and infusions, 3) Follow-up after infusions.
* Pre-infusion evaluation: Routine blood tests will be performed on both the participant and donor. The participant will undergo a bone marrow aspirate and biopsy if this has not been recently performed. During this time, additional standard blood tests and/or radiology tests may be done to fully determine the extent of the cancer.
* Cell Collections: About 2-3 weeks before the infusion date, the donor will undergo one or two white blood cell collection procedures called leukopheresis. The cells collected from the first leukopheresis will be sent to the laboratory where a portion will be used to cultivate dendritic cells, and the remaining lymphocytes will be set aside for the DLI. If the number of cells collected at the first leukopheresis is insufficient, the donor will undergo a second leukopheresis procedure 7-10 days later.
* Infusions: We plan to administer the dendritic cells and donor lymphocytes separately in the outpatient clinic. The dendritic cells will be given first, followed by the DLI one to two days later.
* Follow-up after infusions: After completion of both the donor DC and DLI, participants will be followed closely for the development of side effects and response. They will be evaluated at least once a week, and routine blood tests and physical examination to assess for graft vs. host disease (GvHD) or other side effects will be performed. Additional blood tests will be done after 3, 6, and 10 weeks. At 10 weeks after the lymphocyte infusion, bone marrow aspirate and biopsy will be performed to assess the disease as well as the percentage of bone marrow cells that are derived from the donor. Additional restaging studies will also be performed at 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies who have relapsed after related or unrelated donor hematopoietic stem cell transplantation (e.g. CML, AML, ALL, MDS, NHL, HD, CLL, MM)
* At least two months following hematopoietic stem cell transplantation
* Patients off any systemic immunosuppressive medication for treatment or prevention of GVHD for minimum of 2 weeks prior to initiation of therapy
* 18 years of age or older
* ECOG performance status 0-2
* Donor medically fit to undergo leukapheresis procedure

Exclusion Criteria:

* Relapsed CML in chronic phase
* Prior donor lymphocyte infusion or other immunotherapy treatment within 8 weeks of enrollment
* Clinically significant and active autoimmune disease in donor or patient
* Evidence of active grade II-IV acute GVHD or active extensive chronic GVHD
* Uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-07; Primary Completion 2007-08 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of allogeneic DC in combination with DLI in patents with a relapsed hematologic malignancy following allogeneic hematopoietic stem cell transplantation. | 4 years

SECONDARY OUTCOMES:
To assess clinical response after infusions of donor derived DC and donor lymphocytes
To assess the immunologic impact of infusions of donor derived DC and donor lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Alyea, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts